CLINICAL TRIAL: NCT01595022
Title: A Multi-center, Single-blinded, Randomized, Controlled, Parallel-group Study to Evaluate the Wearing Comfort of Two Different Placebo Intrauterine Systems FR01 and FR20 Compared to a Placebo T-frame Intrauterine System for 3 Cycles in Healthy Women Aged 18-40 Years
Brief Title: FR01 and FR20 IUS (Intrauterine System) Wearing Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13830
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Contraception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flexi ring FR01 (Placebo Comparator)
  Interventions: Drug: Placebo: Flexi ring FR01
- Flexi ring FR20 (Placebo Comparator)
  Interventions: Drug: Placebo: Flexi ring FR20
- Ultra low dose LCS (Placebo Comparator)
  Interventions: Drug: Placebo: Ultra low dose levonorgestrel contraceptive system (LCS)

INTERVENTIONS:
Drug: Placebo: Flexi ring FR01 — Intrauterine device, inserted once for 3 months
  Arms: Flexi ring FR01
Drug: Placebo: Flexi ring FR20 — Intrauterine device, inserted once for 3 months
  Arms: Flexi ring FR20
Drug: Placebo: Ultra low dose levonorgestrel contraceptive system (LCS) — Intrauterine device, inserted once for 3 months
  Arms: Ultra low dose LCS

SUMMARY:
The aim of the study is to evaluate two different placebo intrauterine systems, placebo FR01 and FR20 with different types of inserters, for wearing comfort, insertion/removal ease and pain compared to a placebo T-frame intrauterine system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female subject
* Age 18-40 years (inclusive)
* History of regular cyclic menstrual periods at baseline (cycle length 21 to 35 days)
* Women using any COC (combined oral contraceptive) for contraception with a monthly regimen before the study entry.
* Confirmed uterine sound depth of 6 to 10 cm

Exclusion Criteria:

* Pregnancy or lactation
* Sterilized
* Nulliparous
* Congenital or acquired uterine anomaly
* Vaginal or cesarean delivery within 8 weeks prior to insertion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pelvic pain during the IUS wearing period (wearing comfort) measured by 5-point Likert scale (no pain/mild/moderate/severe/very severe pain) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Finland (4):
  - Helsinki
  - Kuopio
  - Tampere
  - Turku
- Netherlands (3):
  - Den Helder
  - Heerlen
  - Zwijndrecht
- Sweden (3):
  - Örebro
  - Stockholm
  - Uppsala